CLINICAL TRIAL: NCT02784288
Title: Phase II Treatment Stratification Trial Using Neck Dissection-Driven Selection to Improve Quality of Life for Low Risk Patients With HPV+ Oropharyngeal Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.126; HUM00105447 (Other: University of Michigan)
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Oropharyngeal Squamous Cell Cancer
Keywords: head and neck neoplasms; HPV; human papilloma virus; de-escalation; low-risk; oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Neck Dissection; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neck Dissection (Experimental): Patients undergo up-front neck dissection of the cervical lymph nodes to determine stratification into one of three standard-of-care treatment groups: transoral surgery of the primary site, radiation or chemoradiation.
  Interventions: Procedure: Neck Dissection; Procedure: Standard-of-Care (SOC) Transoral Surgery of Primary Site; Radiation: SOC Radiation; Drug: SOC Carboplatin; Drug: SOC Paclitaxel; Procedure: Videofluoroscopy

INTERVENTIONS:
Procedure: Neck Dissection — All patients will undergo neck dissection of the cervical lymph nodes
Procedure: Standard-of-Care (SOC) Transoral Surgery of Primary Site — Patients with a single lymph node that measures less than six centimeters, have no extracapsular extension in the lymph node, and have no perineural or perivascular invasion of the primary biopsy will undergo transoral surgery of the primary site.
Radiation: SOC Radiation — Patients who have 2 positive nodes with no extracapsular extension, or have perineural or perivascular invasion of the primary biopsy will undergo radiation.
Drug: SOC Carboplatin — Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation (Radiation, Carboplatin and Paclitaxel).
Drug: SOC Paclitaxel — Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation (Radiation, Carboplatin and Paclitaxel).
Procedure: Videofluoroscopy — All patients undergo a videofluoroscopy procedure one year after completion of therapy to assess swallowing function.

SUMMARY:
Investigators will determine whether a treatment paradigm of up-front neck dissection, to more accurately pathologically stage patients, minimizing the number of treatment modalities in patients with low risk oropharyngeal squamous cell carcinoma, can improve quality of life.

DETAILED DESCRIPTION:
After enrollment, all patients will undergo neck dissection and primary site biopsy. Pathology will be reviewed, and patients will proceed into one of three standard-of-care (SOC) treatment groups. The treatments themselves are not the focus of this study; the focus of this study is quality of life in this population, after a pathology-based treatment plan, to assess the utility of the investigational "neck dissection first" paradigm. The SOC treatment plans are as follows:

1. Patients with a single lymph node that measures less than six centimeters, have no extracapsular extension in the lymph node, and have no perineural or perivascular invasion of the primary biopsy will undergo transoral surgery of the primary site.
2. Patients who have 2 positive nodes with no extracapsular extension, or have perineural or perivascular invasion of the primary biopsy will undergo radiation.
3. Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation.

After completion of therapy (surgical, radiation, or combined modality) patients will be followed closely on an outpatient basis including regular exams, quality of life questionnaires, and interval surveillance imaging as clinically indicated. Swallowing function will also be addressed by videofluoroscopy one year after completion of therapy. Blood/plasma and oral rinses for correlative studies will be collected at 3-month intervals during 3 years of follow up.

This study was initially registered as if it were an inter-group comparison; however, the original and consistent intent has been to determine whether a treatment paradigm of neck dissection guided staging as a whole can minimize the number of standard treatment methods used, leading to improved quality of life in low risk patients with HPV+ oropharyngeal squamous cell cancer. Though certain groups are expected to need multimodal definitive treatment downstream of the experimental "neck dissection first" paradigm, the population must be assessed as one group in this trial to assess the utility of the paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, previously untreated, p16-positive oropharyngeal squamous cell carcinoma
* Patients must have pretreatment neck and chest imaging
* Tumors must be potentially surgically resectable via a transoral approach, at the discretion of the treating surgeon
* Patients with T stage T1-3
* Patients with N stage N0-N2c
* ECOG (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.) Performance status 0-2
* Patients are adults (Age >18)
* Patients must agree to biospecimen submission for tissue and serum processing and storage for secondary biomarker studies
* Patients must give documented informed consent to participate in this study.
* Patients must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of chemoradiation (treatment) and for 3 months after discontinuing treatment. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to starting treatment.
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 30 days after study treatment. Women not of childbearing potential will be defined as all women older than age 50 and anovulatory for 12 months.
* Sexually active males must use a condom during intercourse while receiving chemoradiation and for 90 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. Likewise, male subjects should not donate sperm during the time they are receiving chemoradiation and for 90 days after stopping treatment.

Exclusion Criteria:

* Prior head and neck radiation or prior chemotherapy for HNSCC (Head and Neck Squamous Cell Carcinoma)
* Patients with T4 disease
* Patients with N3 disease
* FNA evidence of squamous cell carcinoma involving 3 or more lymph nodes
* Patients with matted lymph nodes, defined as three nodes abutting one another with loss of intervening fat plane that is a replaced with radiologic evidence of extracapsular spread
* Patients with an outside primary site biopsy showing perineural or perivascular invasion
* Documented evidence of distant metastases.
* Active infection
* Patients residing in prison.
* Age < 18 years
* Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Unstable angina or a history of myocardial ischemia within prior 6 months
* Patients with any of the following laboratory values at baseline:

  * Absolute neutrophil count (ANC) < 1,000/mm3
  * Platelets < 75,000/mm3
  * Hemoglobin < 9.0 gm/dL
  * Calculated or measured creatinine clearance (method determined by the prescribing physicians) < 50 ml/min
  * Bilirubin > 1.5 x ULN (Upper Limit of Normal), except for patients with known Gilbert syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN
  * Aspartate transaminase (AST) > 3.0 x ULN
  * Alanine transaminase (ALT) > 3.0 x ULN
* Pregnancy or breastfeeding female.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swiecicki, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients consented only 34 enrolled and started on treatment
Period: Overall Study
Arm/Group | Neck Dissection
Started | 34
Completed | 33
Not Completed | 1
Not completed — Patients neck dissection had spillage and therefore needed to come off protocol | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neck Dissection
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 60 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Quality of Life (QOL) From Baseline to 12 Months Post Treatment
Description: Four QOL instruments will be administered: the University of Washington Quality of Life (UWQOL), University of Michigan Head and Neck Quality of Life Instrument (HN-QOL), the University of Michigan Voice Related Quality of Life Measure (V-RQOL), and the FACT Head and Neck (version 4) (FACT H&N). Results of each of the 4 surveys will be reported in separate rows in the results table. The difference in scores from baseline to 12 months after completion of study treatment is calculated for each participant, with the median across all participants reported for each survey. Higher scores indicate better QOLs.
  Range for Questionnaires:
  HN QOLs: -100 to +100 VR QOLs: -100 to +100 UW QOLs: -100 to +100 FACTHN Physical: -28 to +28 FACTHN Social: -28 to +28 FACTHN Emotional: -24 to +24 FACTHN Functional: -28 to +28 FACTHN subscale: -40 to +40 FACTHN Total: -148 to +148
Time Frame: Baseline to 12 Months post-treatment (up to approximately 15 months post neck dissection).
Population: only 19 patients, out of 34, were compliant in completing the 12 month QOLs.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Neck Dissection
Number analyzed (Participants) | 19
score on a scale
  HN-QOL: Eating | -4.2 [-37.5 to 29.2]
  HN-QOL: Speech | 0 [-37.5 to 25]
  HN-QOL: Pain | 6.3 [-18.8 to 37.5]
  HN-QOL: Emotion | 10.7 [-3.6 to 25]
  UW-QOL: Pain_general | 0 [-40 to 0]
  UW-QOL: Pain_mouth | 0 [-30 to 10]
  UW-QOL: Pain_throat | -10 [-20 to 10]
  UW-QOL: Disfigurement | 0 [-10 to 20]
  UW-QOL: Activity | 0 [-10 to 10]
  UW-QOL: Recreation | 0 [-10 to 10]
  UW-QOL: Employment: number analyzed (Participants) | 17
  UW-QOL: Employment | 0 [0 to 20]
  UW-QOL: Chewing | 0 [-20 to 10]
  UW-QOL: Swallowing | 0 [-30 to 10]
  UW-QOL: Saliva amount | 10 [0 to 40]
  UW-QOL: Saliva consistency: number analyzed (Participants) | 18
  UW-QOL: Saliva consistency | 0 [-20 to 10]
  UW-QOL: Taste | 10 [-10 to 30]
  UW-QOL: Speech | 0 [-10 to 10]
  UW-QOL: Mucus amount | 0 [-30 to 20]
  UW-QOL: Mucus consistency | 0 [-20 to 20]
  V-RQOL: Physical: number analyzed (Participants) | 18
  V-RQOL: Physical | 0 [-0.2 to 0.04]
  V-RQOL: Emotional: number analyzed (Participants) | 18
  V-RQOL: Emotional | 0 [-0.06 to 0]
  V-RQOL: Total: number analyzed (Participants) | 18
  V-RQOL: Total | 0 [-0.1 to 0.03]
  FACT H&N: Physical Well Being | 1 [-6 to 7]
  FACT H&N: Social Well Being | 0 [-7.5 to 5]
  FACT H&N: Emotional Well Being | 3 [-4 to 6]
  FACT H&N: Functional Well Being | 0 [-9 to 7]
  FACT H&N: HN subscale | -1 [-12 to 12]
  FACT H&N: Total | 4 [-21 to 19]

2. Secondary Outcome: Impact of Neck Dissection on Shoulder Function Using the Neck Dissection Impairment Index
Description: The neck dissection impairment index will be scored and summarized for all patients who receive neck dissection.
  Scores ranging from 0-100 with higher scores indicating better function
Time Frame: 2 years post-treatment (up to approximately 27 months post neck dissection)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Neck Dissection
Number analyzed (Participants) | 20
score on a scale | 98 [78 to 100]

3. Secondary Outcome: Median Change in Quality of Life (QOL) From Baseline to 24 Months Post Treatment
Description: Four QOL instruments will be administered: the University of Washington Quality of Life (UWQOL), University of Michigan Head and Neck Quality of Life Instrument (HN-QOL), the University of Michigan Voice Related Quality of Life Measure (V-RQOL), and the FACT Head and Neck (version 4) (FACT H&N). Results of each of the 4 surveys will be reported in separate rows in the results table. The difference in scores from baseline to 24 months after completion of study treatment is calculated for each participant, with the median across all participants reported for each survey. Higher scores indicate better QOLs.
  Range for Questionnaires:
  HN QOLs: -100 to +100 VR QOLs: -100 to +100 UW QOLs: -100 to +100 FACTHN Physical: -28 to +28 FACTHN Social: -28 to +28 FACTHN Emotional: -24 to +24 FACTHN Functional: -28 to +28 FACTHN subscale: -40 to +40 FACTHN Total: -148 to +148
Time Frame: 2 years post-treatment (up to approximately 27 months post neck dissection)
Population: only 19 patients, out of 34, were compliant in completing the 24 month QOLs
Measure: Median (Full Range); unit: score on a scale
Groups:
- Neck Dissection: Patients underwent up-front neck dissection of the cervical lymph nodes to determine stratification into one of three standard-of-care treatment groups: transoral surgery of the primary site, radiation or chemoradiation.
  Neck Dissection: All patients will undergo neck dissection of the cervical lymph nodes
  Standard-of-Care (SOC) Transoral Surgery of Primary Site: Patients with a single lymph node that measures less than six centimeters, have no extracapsular extension in the lymph node, and have no perineural or perivascular invasion of the primary biopsy will undergo transoral surgery of the primary site.
  SOC Radiation: Patients who have 2 positive nodes with no extracapsular extension, or have perineural or perivascular invasion of the primary biopsy will undergo radiation.
  SOC Carboplatin: Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation (Radiation, Carboplatin and Paclitaxel).
  SOC Paclitaxel: Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation (Radiation, Carboplatin and Paclitaxel).
  Videofluoroscopy: All patients undergo a videofluoroscopy procedure one year after completion of therapy to assess swallowing function.
Arm/Group | Neck Dissection
Number analyzed (Participants) | 19
score on a scale
  HN-QOL- Eating | 0.0 [-41.7 to 29.2]
  HN-QOL- Speech | 0.0 [-12.5 to 25.0]
  HN-QOL- Pain | 6.3 [-18.8 to 31.3]
  HN-QOL- Emotion | 10.7 [-3.6 to 28.6]
  UWQOL-Pain_General | -10 [-30 to 10]
  UWQOL- Pain_Mouth | 0 [-20 to 10]
  UWQOL- Pain_throat | -10 [-20 to 10]
  UWQOL- Disfigurement | 0 [-10 to 20]
  UWQOL- activity | 0 [-10 to 10]
  UWQOL-Recreation | 0 [-10 to 10]
  UWQOL- Employment | 0 [-30 to 40]
  UWQOL- Chewing | 0 [-20 to 30]
  UWQOL- Swallowing | 0 [-40 to 10]
  UWQOL- Saliva amount | 10 [0 to 40]
  UWQOL- Saliva consistency: number analyzed (Participants) | 18
  UWQOL- Saliva consistency | 0 [-10 to 40]
  UWQOL- Taste | 0 [-30 to 20]
  UWQOL- Speech | 0 [-10 to 20]
  UWQOL- Mucus amount | 0 [-40 to 20]
  UWQOL- Mucus consistency | 0 [-40 to 20]
  V-RQOL- Physical: number analyzed (Participants) | 17
  V-RQOL- Physical | 0 [-0.1 to 0.10]
  V-RQOL- Emotional: number analyzed (Participants) | 17
  V-RQOL- Emotional | 0 [-0.3 to 0]
  V-RQOL- Total: number analyzed (Participants) | 17
  V-RQOL- Total | 0 [-0.2 to 0.06]
  FACT H&N- Physical well being: number analyzed (Participants) | 17
  FACT H&N- Physical well being | 0 [-6 to 6]
  FACT H&N- Social well being: number analyzed (Participants) | 17
  FACT H&N- Social well being | 0 [-8.5 to 9.3]
  FACT H&N- Emotional well being: number analyzed (Participants) | 17
  FACT H&N- Emotional well being | 2 [-4 to 5]
  FACT H&N- Functional well being: number analyzed (Participants) | 17
  FACT H&N- Functional well being | 0 [-7 to 11]
  FACT H&N- HN subscale: number analyzed (Participants) | 17
  FACT H&N- HN subscale | 2 [-17 to 11]
  FACT H&N- total FACTHN: number analyzed (Participants) | 17
  FACT H&N- total FACTHN | 1 [-20 to 31.3]

4. Secondary Outcome: Disease Specific Survival (DSS)
Description: Proportion of patients alive at 3 years from date of neck dissection. Death from OPSCC (Oropharyngeal Squamous Cell Cancer) will be considered an event for DSS. Death from other causes will be censored at time of death.
Time Frame: 3 Years
Measure: Number; unit: percentage of participants
Arm/Group | Neck Dissection
Number analyzed (Participants) | 33
percentage of participants | 100

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Proportion of patients alive and free of disease persistence, progression or recurrence at 3 years from the date of completion of study treatment. Persistent disease at completion of treatment, post-treatment recurrence or disease specific death will be defined events for progression free survival (PFS).
Time Frame: 3 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neck Dissection
Number analyzed (Participants) | 33
percentage of participants | 97 [76 to 99]

6. Secondary Outcome: Overall Survival (OS)
Description: Proportion of patients alive at 3 years from date of neck dissection. Death from any cause will be considered an event for overall survival.
Time Frame: 3 Years
Measure: Number; unit: Percent of Patients
Arm/Group | Neck Dissection
Number analyzed (Participants) | 33
Percent of Patients | 100

ADVERSE EVENTS:
Time Frame: up to 12 months post treatment for Adverse Events, Serious Adverse Events up to 4 weeks post treatment, All-Cause Mortality assessed up to 3 years
Groups:
- Neck Dissection: Patients undergo up-front neck dissection of the cervical lymph nodes to determine stratification into one of three standard-of-care treatment groups: transoral surgery of the primary site, radiation or chemoradiation:
  Neck Dissection: All patients will undergo neck dissection of the cervical lymph nodes
  SOC Transoral Surgery of Primary Site: Patients with a single lymph node that measures less than six centimeters, have no extracapsular extension in the lymph node, and have no perineural or perivascular invasion of the primary biopsy will undergo transoral surgery of the primary site.
  SOC Radiation: Patients who have 2 positive nodes with no extracapsular extension, or have perineural or perivascular invasion of the primary biopsy will undergo radiation.
  SOC Carboplatin: Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation.
  SOC Paclitaxel: Patients who have extracapsular extension in any number of lymph nodes or in those patients in whom negative margins are unable to be obtained after the completion of transoral surgery will undergo chemoradiation.
  Videofluoroscopy: All patients undergo a videofluoroscopy procedure one year after completion of therapy to assess swallowing function.
  All patients, regardless of intervention were combined into one arm for analysis
Arm/Group | Neck Dissection
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neck Dissection (N=34)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral Hemorrhage (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neck Dissection (N=34)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders- Other (Cardiac disorders) | 1 (1)
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (9)
Depression (Psychiatric disorders) | 4 (4)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 20 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 19 (34)
Dysphagia (Gastrointestinal disorders) | 17 (29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 5 (8)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 6 (10)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Facial pain (General disorders) | 2 (2)
Fatigue (General disorders) | 14 (22)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions- Other (General disorders) | 10 (18)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (6)
Hearing impaired (Ear and labyrinth disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 6 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 4 (5)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Lymphedema (Vascular disorders) | 6 (6)
Lymphocyte count decreased (Investigations) | 3 (7)
Meningismus (Nervous system disorders) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (20)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 14 (21)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 14 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (3)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Testicular disorder (Reproductive system and breast disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 6 (6)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 14 (14)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT02784288/Prot_SAP_ICF_000.pdf